CLINICAL TRIAL: NCT04324528
Title: Cytokine Adsorption in Severe COVID-19 Pneumonia Requiring Extracorporeal Membrane Oxygenation
Acronym: CYCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Alexander Supady (Other)
Responsible Party: Sponsor-Investigator, Dr. Alexander Supady, Attending Physician - Oberarzt, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYCOV
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus; COVID-19; SARS-CoV Infection; Respiratory Failure; Cytokine Storm
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome; Respiratory Insufficiency; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: randomized controlled trial examining COVID-patients requiring vv-ECMO therapy (+/- cytokine adsorption)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vv-ECMO + cytokine adsorption (Experimental): after indication of treatment with vv-ECMO in acute respiratory failure in COVID-19-disease, patients will additionally receive cytokine adsorption using a Cytosorb adsorber
  Interventions: Device: vv-ECMO + cytokine adsorption (Cytosorb adsorber)
- control-arm: vv-ECMO (no cytokine adsorption) (Other): treatment with vv-ECMO in acute respiratory failure in COVID-19-disease (standard treatment without additional cytokine adsorption)
  Interventions: Device: vv-ECMO only (no cytokine adsorption)

INTERVENTIONS:
Device: vv-ECMO + cytokine adsorption (Cytosorb adsorber) — in COVID-19-diseased vv-ECMO patients additional treatment with cytokine adsorption using a Cytosorb adsorber will be randomized (vs. control group)
  Arms: vv-ECMO + cytokine adsorption
Device: vv-ECMO only (no cytokine adsorption) — COVID-19-diseased treated with vv-ECMO
  Arms: control-arm: vv-ECMO (no cytokine adsorption)

SUMMARY:
In December 2019 in the city of Wuhan in China, a series of patients with unclear pneumonia was noticed, some of whom have died of it. In virological analyses of samples from the patients' deep respiratory tract, a novel coronavirus was isolated (SARS-CoV-2). The disease spread rapidly in the city of Wuhan at the beginning of 2020 and soon beyond in China and, in the coming weeks, around the world.

Initial studies described numerous severe courses, particularly those associated with increased patient age and previous cardiovascular, metabolic and respiratory diseases. A small number of the particularly severely ill patients required not only highly invasive ventilation therapy but also extracorporeal membrane oxygenation (vv-ECMO) to supply the patient's blood with sufficient oxygen.

Even under maximum intensive care treatment, a very high mortality rate of approximately 80-100% was observed in this patient group. In addition, high levels of interleukin-6 (IL-6) could be detected in the blood of these severely ill patients, which in turn were associated with poor outcome.

From experience in the therapy of severely ill patients with severe infections and respiratory failure, we know that treatment with a CytoSorb® adsorber can lead to a reduction of the circulating pro- and anti-inflammatory cytokines and thus improve the course of the disease and the outcome of the patients.

Our primary goal is to investigate the efficacy of treatment with a CytoSorb® adsorber in patients with severe COVID-19 disease requiring venous ECMO over 72 hours after initiation of ECMO. The primary endpoint is the reduction of plasma interleukin-6 levels 72 hours after initiation of ECMO support. As secondary endpoints we investigate 30-day survival, vasopressor and volume requirements, lactate in terms of lactate and platelet function. As safety variables, we further investigate the levels of the applied antibiotics (usually ampicillin and sulbactam).

DETAILED DESCRIPTION:
In December 2019, a series of unexplained cases of pneumonia in the city of Wuhan in China has come to light. In virological analyses of samples from the patients' deep respiratory tract, a novel coronavirus was isolated (first named 2019-nCoV, then SARS-CoV-2). The disease spread rapidly in the city of Wuhan in early 2020 and soon beyond. On 30 January 2020, the Director-General of the World Health Organization (WHO) declared the outbreak a public health emergency of international concern, and on 11 March 2020, the World Health Organization declared the virus a pandemic.

In humans, an infection with the virus can cause respiratory infections and even very severe pneumonia, which often ends fatally, especially in old and previously ill patients. Due to the novelty of the virus, the data basis for therapy is very limited. To date, there are no clinical data for an effective specific therapy, nor is there a vaccination against the virus available, so that therapy, especially intensive care treatment for very severe cases, must concentrate only on supportive treatment of lung failure and other complications.

The virus is very contagious and infection results in a relevant number of deaths. Due to very uncertain data on the spread of the virus in the population, it is difficult to estimate the mortality rate - case mortality is about 4% based on known case numbers.

In reports on the treatment of the first cases in Wuhan (Hubei Province, China) in January 2020, the need for intensive care treatment is described for about a quarter of the inpatient cases, 10-17% had to be ventilated invasively, and venous extracorporeal membrane oxygenation (vv-ECMO) was necessary in 2-4% of the inpatient cases. Patients requiring ECMO have an extremely high mortality rate of 83-100% in the studies described so far.

In severe cases a pronounced release of vasoactive cytokines was repeatedly observed. Excessive release of these vasoactive mediators ("cytokine storm") can result in pronounced vasodilatation and membrane leakage, which can ultimately lead to severe vasoplegic shock that is difficult to control. Ruan et al. and Zhou et al. have identified high interleukin 6 (IL-6) levels as a potential predictor of a fatal outcome when compared between survivors and patients who died of COVID-19 disease.

IL-6 is also an important factor in the pathophysiology of severe septic shock and excessive immune response in hemophagocytic lymphohistiocytosis (HLH) - for both indications has been shown, that the extracorporeal adsorption of IL-6 and other vasoactive substances in a CytoSorb® adsorber (CytoSorbents Corporation, Monmouth Junction, NJ, USA) leads to a significant reduction of these cytokines in the patient blood. Clinical experience and (previously unpublished) data from our monocentric registry study show that cytokine adsorption in a CytoSorb® Adsorber can also be safely integrated into a vv-ECMO system.

The aim of the study is to investigate the influence of extracorporeal cytokine adsorption on humoral inflammation parameters and patient survival under controlled conditions in patients with severe COVID-19 disease requiring extracorporeal membrane oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2-infection with COVID-pneumonia
* vv-ECMO therapy

Exclusion Criteria:

* pregnancy, breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
interleukin-6 (IL-6) level after 72 hours | 72 hours
  measurement of IL-6 levels in patient blood after 72 hours of cytokine adsorption (in relation to level before initiation of cytokine adsorption)

SECONDARY OUTCOMES:
30-day-survival | 72 hours
  survival after 30 days
vasopressor dosage | 72 hours
  needed dosage of norepinephrine and other vasopressors
fluid balance | 72 hours
  fluid balance levels during cytokine adsorption
lactate | 72 hours
  serum-lactate levels during cytokine adsorption

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Supady, Dr., MPH, Principal Investigator — University Clinic Freiburg
Locations (1):
- University Clinic Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Supady A, Weber E, Rieder M, Lother A, Niklaus T, Zahn T, Frech F, Muller S, Kuhl M, Benk C, Maier S, Trummer G, Flugler A, Kruger K, Sekandarzad A, Stachon P, Zotzmann V, Bode C, Biever PM, Staudacher D, Wengenmayer T, Graf E, Duerschmied D. Cytokine adsorption in patients with severe COVID-19 pneumonia requiring extracorporeal membrane oxygenation (CYCOV): a single centre, open-label, randomised, controlled trial. Lancet Respir Med. 2021 Jul;9(7):755-762. doi: 10.1016/S2213-2600(21)00177-6. Epub 2021 May 14. PMID 34000236